CLINICAL TRIAL: NCT05254418
Title: Effects of Glucagon-Like Peptide-1 Agonists on Metabolism and Ectopic Fat Deposition in Chronic Kidney Disease: A Pilot and Feasibility Study
Brief Title: Effects of GLP1-RA on Ectopic Fat Deposition in Chronic Kidney Disease
Acronym: GLIMP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: VA Tennessee Valley Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alp Ikizler, Catherine McLaughlin Hakim Chair in Vascular Biology, Professor of Medicine, Director, Division of Nephrology and Hypertension, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 220057
Record Dates: First submitted 2022-02-01; First posted 2022-02-24 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease; Intermuscular fat deposition; Glucagon-like peptide-1 agonist; Insulin resistance; Mitochondrial function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Insulin Resistance | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- dulagutide arm (Experimental): Patient will receive 1.5 mg injections per week for 12 weeks.
  Interventions: Drug: dulaglutide injection

INTERVENTIONS:
Drug: dulaglutide injection — All participants will undergo a 4-week run-in phase followed by 12 weeks of treatment (dulaglutide 1.5 mg/wk), followed by 4 weeks of follow up after discontinuing the study medication

SUMMARY:
Chronic kidney disease (CKD) is a burden of morbidity and mortality. Increased protein breakdown in skeletal muscle (wasting) and ectopic fat deposition are important determinants of poor clinical outcome in patient with CKD. Insulin resistance plays a critical role in skeletal muscle wasting and ectopic fat deposition. Glucagon-like peptide-1 receptor agonists (GLP-1RA) decrease ectopic fat deposition in patients with type 2 diabetes, prediabetes, obese and overweight subjects.

The influence of GLP-1RA on ectopic fat deposition in CKD patients in unknown. The investigators' will test the hypothesis that GLP-1RA decreases intermuscular (ectopic) fat deposition in patients with stage 3-4 CKD. The investigators' will do so by addressing the following specific aims:

Specific Aim 1: To test the hypothesis that GLP-1RA decreases intermuscular fat deposition in patients with stage 3-4 CKD.

Specific Aim 2: To test the hypothesis that GLP-1RA improves skeletal muscle mitochondrial function in patients with stage 3-4 CKD.

Specific Aim 3: To test the hypothesis that GLP-1RA improves physical performance in patients with stage 3-4 CKD.

Specific Aim 4: To test the safety and feasibility of 12 weeks of dulaglutide 1.5 mg/wk administration as an adjunct therapy to the standard care of patients with stage 3-4 CKD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage 3-4 CKD (eGFR 15-59 ml/min/1/73 m2)
2. Age ≥ 18 years and ≤75 years

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus
2. Patients with T2D who are on insulin therapy or who started a new antidiabetic medication within 1 month prior to study or who received incretin-based therapy within 3 months prior to study
3. BMI <25 kg/m2, BMI >40 kg/m2
4. HbA1c>8% measured within 1 month prior to study, or a history of hypoglycemic episode within 1 year prior to study, or a history of diabetic ketoacidosis
5. Uncontrolled hypertension (>200/100 mmHg) despite optimal antihypertensive therapy
6. Arrythmia, heart failure (NYHA class III-IV), valve disease or heart diseases other than coronary artery disease
7. History of major gastrointestinal surgery, inflammatory bowel disease, pancreatitis or cholelithiasis
8. Personal or family history of medullary thyroid cancer, or personal history of Multiple Endocrine Neoplasia (MEN)-2
9. Pregnancy, breast feeding or intention to become pregnant
10. Previous renal transplantation
11. Acute or chronic infectious diseases
12. Cancer or chemotherapy within 3 years prior to study
13. Treatment with systemic corticosteroids within 3 months prior to study
14. Known or suspected allergy to dulaglutide
15. Claustrophobia or other contraindications for magnetic resonance imaging

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dulagutide Arm
Started | 7
Completed | 5
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dulagutide Arm
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Changes in Intermuscular Fat Deposition as Assessed by Magnetic Resonance Imaging (MRI).
Description: Sequential MRI will be performed during the run-in phase, at the beginning and end of the dulaglutide treatment and at the end of the observational follow up period. Intermuscular fat will be calculated as the ratio between intermuscular fat and muscle volumes in the mid-thigh region. Changes in intermuscular fat deposition will be calculated. the reported value is the difference between the end of study and baseline values (end of study minus baseline). A negative value will reflect a decrease in IMAT.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: fat/muscle ratio
Arm/Group | Dulagutide Arm
Number analyzed (Participants) | 7
fat/muscle ratio | -0.009 (0.0526)

2. Primary Outcome: Changes in Skeletal Muscle Mitochondrial Function as Assessed by Phosphocreatine Recovery Time Constant by 31P Magnetic Resonance Spectroscopy (31P-MRS).
Description: Sequential 31P-MRS, a gold standard technique for muscle mitochondrial function assessment, will be performed during the run-in phase, at the beginning and end of the dulaglutide treatment and at the end of the observational follow up period. Changes in phosphocreatine recovery time constant will be assessed.
Time Frame: 16 weeks
Population: MRS data could not be reported as the required acquisition was not completed. The estimated scan duration exceeded two hours, and there was insufficient time within the reserved scan slot to perform this portion. Additionally, the patients were unable to tolerate the prone position for such an extended period, which ultimately prevented the collection of data necessary for MRS analysis.
Groups:
- Intervention: Patient will receive 1.5 mg injections per week for 12 weeks
Arm/Group | Intervention
Number analyzed (Participants) | 0

3. Primary Outcome: Changes in Physical Performance as Assessed by Systemic Physical Performance Battery Test
Description: Systemic physical performance battery test will be performed at the beginning and end of the dulaglutide treatment period. Changes will be assessed. The total score that will be reported is calculated by adding scores obtained from Balance test, Gait speed test and Chair stand test scores. The score for the primary outcome will be the difference between baseline and end of study.
  The SPPB total score ranges from 0 (worst performance) to 12 points (best performance) and categorically evaluates performance in the tests using three or four classes of scores: three classes: 0-6 points (poor performance), 7-9 points (moderate performance), and 10-12 points (good performance); or four classes: 0-3 points (disability/very poor performance), 4-6 points (poor performance), 7-9 points (moderate performance), and 10-12 points (good performance)
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulagutide Arm
Number analyzed (Participants) | 7
score on a scale | 0 (2.24)

4. Primary Outcome: Safety and Feasibility of Dulaglutide Treatment as Evaluated by Subject Interview, Continuous Glucose Monitoring, Adverse Events (AE), Laboratory Tests, Vital Signs, ECG & Allergic/Hypersensitivity Reactions.
Description: An AE will be defined as any undesirable medical event occurring to a subject in a clinical trial, whether it is related to the study agent. All adverse events will be graded as follows: 0 = No adverse events or within normal limits; 1 = Mild-did not require treatment; 2 = Moderate resolved with treatment; 3 = Severe-required professional medical attention; 4 = Life-threatening or disabling; 5 = Death.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dulagutide Arm
Number analyzed (Participants) | 7
Participants | 2

ADVERSE EVENTS:
Time Frame: 16 weeks: 12 weeks while the patient is on the medication and 4 weeks of follow up after the study is completed. There is only one arm in this study.
Groups:
- Run-in-Period: Patient will undergo a 4-week run in phase before starting the intervention.
- Dulagutide Arm: Patient will receive 1.5 mg injections per week for 12 weeks.
  dulaglutide injection: The intervention will start at the beginning of the Treatment Phase and will continue for12 weeks of treatment.
- Follow-up: Patients will undergo a 4 week follow up phase after the intervention and before ending the study.
Arm/Group | Run-in-Period | Dulagutide Arm | Follow-up
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 2/7 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in-Period (N=7) | Dulagutide Arm (N=7) | Follow-up (N=7)
nausea (Gastrointestinal disorders) | NA | 1 (1) | NA
local injection site erythema (Skin and subcutaneous tissue disorders) | NA | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT05254418/Prot_002.pdf
  • Statistical Analysis Plan (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT05254418/SAP_003.pdf